CLINICAL TRIAL: NCT03267017
Title: Correlation Between Respiratory Variability of R-R Intervals and in Invasive Systolic Blood Pressure During Changes in Posture and Positive End Expiratory Pressure
Brief Title: Correlation Between Respiratory Variability of R-R Intervals and Systolic Pressure Variability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Amit Lehavi MD FANZCA, Director of Pediatric Anesthesia, Rambam Health Care Campus
Other Study IDs: RRV PPV
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Heart Rate Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient scheduled for surgery under general anesthesia
  Interventions: Other: posture changes

INTERVENTIONS:
Other: posture changes — Following induction of general anesthesia and initiation of positive pressure ventilation, patients will be tilted 15 degrees head up for 5 minutes with positive end expiratory pressure of 8 cm H2O, and then 15 degrees head down for 5 minutes with positive end expiratory pressure of 3 cm H2O

SUMMARY:
This prospective study is designed to assess and quantify the correlation between respiratory changes in R-R interval and the respiratory changed in invasive systolic blood pressure in ventilated patients during changes in posture and peak end expiratory pressure (PEEP) and following a fluid bolus

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Scheduled for surgery under general anesthesia requiring invasive blood pressure monitoring

Exclusion Criteria:

* Heart Rate other than sinus
* Cardiac Pacemaker Status
* Transplanted Heart

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Statistical Correlation between respiratory variability of R-R interval and systolic blood pressure | From immediately after induction of general anesthesia and mechanical ventilation to 20 minutes later

IPD SHARING:
Plan to Share IPD: No